CLINICAL TRIAL: NCT00960843
Title: A Randomized, Controlled, 6-month Study to Compare the Effects of Volume- and Pressure-guided Adjustments on Weight Loss and Satiety in Patients Implanted With the Swedish Adjustable Gastric Band
Brief Title: Six-month Study to Compare the Effects of Volume- and Pressure-Guided Adjustments on Weight Loss and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-08-0009
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Morbid Obesity
Keywords: Morbid Obesity; Gastric Banding; Bariatric Banding; Swedish Adjustable Gastric Band
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Adjustment Group (Active Comparator): Subject whose band adjustments will be made via conventional standard of care (e.g., volume, hunger).
  Interventions: Other: Conventional Adjustment
- Intraband Pressure Arm (Active Comparator): Subjects whose band adjustments will be guided by intraband pressure readings.
  Interventions: Device: Intraband pressure recording system

INTERVENTIONS:
Device: Intraband pressure recording system — Intraband pressure will be measured by a pressure recording system.
  Arms: Intraband Pressure Arm
Other: Conventional Adjustment — Band adjustments will be made via conventional standard of care (e.g., volume, hunger).
  Arms: Conventional Adjustment Group

SUMMARY:
The purpose of this protocol is to determine how band fill volumes that are based on intraband pressure readings can influence the comfortability of the band and to compare weight loss with this methodology to weight loss with the conventional approach recommended in existing product labeling.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend, follow and give informed consent.
* Be at least 18 years of age at time of trial enrollment.
* Had a pre-implantation BMI between 35 and 55 kg/m2.
* Have received a SAGB VC implant 1) 30-60 days (and not undergone first band adjustment yet)prior to the date of enrollment.
* Willingness to be randomized to intraband-based or conventional adjustments
* Willingness to consent to monthly visits and possible measurements of intraband pressure (requiring access to the injection port).
* Willingness to undergo up to 7 band adjustments within the 6-month period of the study.
* Able to sit approximately at a 90 degree-angle, from the floor, for IBP measurements.
* Willingness to return to office visits around the same time of the first in-study adjustment (plus or minus 2 hours)
* Willingness to consent to a limited UGI series if the investigator suspects the presence of a band-related complication or if the intraband pressure recordings deviate from expected.
* Willingness to refrain from taking medications or supplements indicated for or known to induce weight loss.

Exclusion Criteria:

* Females currently known to be pregnant.
* Ongoing or unresolved band perforation or band leakage.
* Ongoing (unresolved) slippage, erosion, or pouch dilation.
* Documented esophageal dysmotility/dyskinesia.
* Ongoing (unresolved) port obstruction or tube kinking.
* Current injection port infection.
* History of band revision or replacement.
* Previously documented or ongoing esophageal dilatation.
* Any condition that, in the opinion of the Investigator, may jeopardize the subject's well-being or the soundness of this study.
* Current use of medications or supplements indicated for or known to induce weight loss at any point during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Adelaide Bariatric Center, Bedford Park, South Australia, Australia
- OB Klinika, a.s., Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Adjustment Group | Intraband Pressure Arm
Started | 25 | 26
Completed | 23 | 21
Not Completed | 2 | 5
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 0 | 4
Not completed — Repeated needle dislodgment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Adjustment Group | Intraband Pressure Arm | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.93) | 45.1 (12.69) | 46.1 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Czech Republic | 12 | 12 | 24
  Australia | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percent Excess Weight Change at Day 180
Description: Percent Excess Weight Change will be calculated per subject as 100% times the difference between screening and Day 180 visit weight divided by the difference between screening weight and ideal body weight for a given sex and height of a subject. Excess weight is defined as the Screening Weight minus the ideal body weight. Ideal body weight is taken from the 1983 Metropolitan Life using the upper limit value of the medium frame range.
Time Frame: Screening to Day 180
Population: Per Protocol Population - all randomized subjects without major protocol violations affecting the validity of pressure or non-pressure data.
Measure: Mean (Standard Deviation); unit: percentage of excess weight at screening
Groups:
- Conventional Arm: Pressure adjustments based on recommendations in the approved label for the Swedish Adjustable Gastric band
- Intraband Pressure Arm: Pressure adjustments based on protocol instructions regarding intraband pressure measurements
Arm/Group | Conventional Arm | Intraband Pressure Arm
Number analyzed (Participants) | 10 | 11
percentage of excess weight at screening | -13.2 (11.1) | -24.2 (17.5)
Statistical Analysis 1: Comparison: Conventional Arm vs Intraband Pressure Arm; Null hypothesis was no difference between arms. Original power calculation specified 24 per group and this was achieved under initial randomization. However, due to failure to follow protocol specified adjustment criteria, pressure and weight data from one site had to be excluded; Test type: Superiority or Other; p = 0.0520, t-test, 2 sided

2. Secondary Outcome: Mean Static Intraband Pressure at Day 180
Description: Mean static Intraband Pressure will be automatically calculated by the Pressure Recording System as the sum of all pressure points divided by the number of seconds X 10 (10Hz data acquisition)
Time Frame: Day 180
Population: Per Protocol population. Note, one subject in the Intraband pressure arm did not provide static intraband pressure measurements at Day 180 and is thus excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Conventional Arm | Intraband Pressure Arm
Number analyzed (Participants) | 10 | 10
mmHg | 0.7 (7.03) | 15.8 (17.82)
Statistical Analysis 1: Comparison: Conventional Arm vs Intraband Pressure Arm; Test type: Superiority or Other; p = 0.0225, t-test, 2 sided

3. Secondary Outcome: Rate of Weight Loss kg/wk at Day 180
Description: Rate of weight loss = (screening weight (kg) - weight at Day 180 visit (kg)) / (number of days between screening and Day 180 visit / 7).
Time Frame: Screening to Day 180
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: kg/week
Arm/Group | Conventional Arm | Intraband Pressure Arm
Number analyzed (Participants) | 10 | 11
kg/week | 0.18 (0.10) | 0.43 (0.32)
Statistical Analysis 1: Comparison: Conventional Arm vs Intraband Pressure Arm; Test type: Superiority or Other; p = 0.0193, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Conventional Adjustment Group | Intraband Pressure Arm
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/26
Other Adverse Events (participants affected / at risk) | 6/25 | 11/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Adjustment Group (N=25) | Intraband Pressure Arm (N=26)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Adjustment Group (N=25) | Intraband Pressure Arm (N=26)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2) | 3 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (4)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 10 (13)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less